CLINICAL TRIAL: NCT05038761
Title: A Prospective Observational Study to Evaluate the Effectiveness and Safety of Cascade® Continuous Glucose Monitoring System in China: A Real World Study
Brief Title: A Study to Learn How Well a Monitoring System Called Continuous Glucose Monitoring (CGM) Which Measures Glucose on an Ongoing Basis Works and How Safe it is in Chinese Patients in Usual Practice
Acronym: CareMins
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21972
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Continuous Glucose Monitoring; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 or type 2 diabetes mellitus participants: Participants will be enrolled after the decision to initiate venous blood glucose testing and Continuous Glucose Monitoring (CGM) system as per investigator's routine treatment practice.
  Interventions: Device: CGM System; Procedure: Standard Venous Blood Glucose Test

INTERVENTIONS:
Device: CGM System — Following the manner of observational study, no intervention will be used for the study.
  Participants will wear the CGM on abdomen or lower area for no longer than 14 days.
Procedure: Standard Venous Blood Glucose Test — Necessary venous blood glucose testing will be performed during the study as clinically required as comparator.

SUMMARY:
Researchers are looking for a better way to help Chinese people who have diabetes to monitor their blood sugar (blood glucose) situation.

There are 2 types of diabetes. In people with type 1 diabetes, the body's immune system attacks and destroys cells in the pancreas that produce a hormone called insulin. In people with type 2 diabetes, the body does not make enough insulin or does not use insulin well. This results in high blood glucose levels. Over time, high blood glucose levels can cause damage to certain parts of the body. These include the eyes, the kidneys, the nerves, and the heart.

There are tests and devices available for doctors and patients to measure blood glucose levels. Repeated measurements of blood glucose levels are needed to see whether the treatments that prevent blood glucose levels from becoming too high work well and to notice when the blood glucose is decreasing too much. Such tracking of the blood glucose is also called blood glucose monitoring. Blood glucose monitoring tests and devices can however be difficult to use, and one test or device may not work for all patients. Researchers think that better monitoring systems would help patients improve the control of their blood glucose levels. This could help stop their diabetes from getting worse.

In this study, the researchers want to learn more about how well a new monitoring system called CGM works in Chinese patients with diabetes. CGM is a continuous glucose monitoring system. It regularly measures the level of glucose in the tissue throughout the day and night. CGM is made up of a small sensor that patients apply in the belly region where it is placed just under the skin, into the so-called subcutaneous tissue. The sensor measures the level of glucose in the fluid that surrounds cells in the subcutaneous tissue. It also has a transmitter which attaches to the sensor and sends via Bluetooth the results to a device, which can instantly display the glucose level. The glucose levels can then be used to adjust the treatment.

The main purpose of this study is to learn how well CGM monitors glucose levels in Chinese patients when used in usual practice. To answer this question, the researchers will compare the glucose levels collected with the CGM monitor to the blood glucose levels collected with another type of monitoring called "venous blood glucose testing". This is where a blood sample is taken from the veins, and then the level of glucose in the blood sample is measured.

The study will include adult Chinese patients who have type 1 or type 2 diabetes and who the study doctors think need to monitor their diabetes using CGM and venous blood glucose testing.

There will be no treatments given as part of this study. The device will be worn up to a maximum of 14 days. The patients will get training on how to use the CGM monitor and will attach it to their belly on Day 1 of the study.

The researchers will then collect the information about their glucose levels. The study doctors will also take blood samples and measure blood glucose levels using venous blood glucose testing. They will compare the glucose levels recorded from the blood samples to the glucose levels recorded by CGM at the closest time points. After wearing CGM for 14 days, the study doctors will remove it from the patients' bellies. About 3 days later, the researchers will call the patients to check if they have any swelling or areas of rash where CGM was worn. The patients may also take photos of the area and send these to the study doctors.

During the study, the study staff will:

* take blood samples as part of the usual care
* compare glucose levels recorded by CGM to the levels recorded from the venous blood glucose tests
* check the skin for any swelling or areas of rash where CGM was worn
* record any instances of CGM errors or alarms for when glucose levels are too high or too low
* check the patients' overall health
* ask the patients about how they are feeling and what medical problems they are having.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male (18 years of age or older)
* Diagnosed with type 1 or type 2 diabetes mellitus
* Decision to initiate venous blood glucose testing and CGM as per investigator's routine treatment practice;
* Signed informed consent

Exclusion Criteria:

* Patients with moderate or more serious anemia defined as hemoglobin < 90g/L
* Patients with moderate or more serious subcutaneous edema: grading can be referred to: mild edema (a visible mild depression of eyelid, soft tissues below the orbit, subcutaneous tissue of the anterior tibia or subcutaneous tissue of the ankle after finger pressure); moderate (all the sparse tissues of the whole body have visible edema with obvious or deeper tissue depressions after finger pressure and slow subsidence); severe (severe edema of tissues all over the body, the skin of the low hanging part of the body is tense and shiny, and there may even be fluid exudation, sometimes accompanied by fluid accumulation in the thoracic cavity, abdominal cavity and sphincter cavity)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and/or male patients with a diagnosis of type 1 or type 2 diabetes mellitus will be enrolled after the decision to initiate venous blood glucose testing and CGM as per investigator's routine treatment practice.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
20/20% agreement rate with reference value | From successful device-wearing to device-removal, up to 14 days
  To compare CGM values with reference venous blood glucose values and to analyze the agreement rate
Percentage of total points found in Zone A +B of Clarke Error Grid | From successful device-wearing to device-removal, up to 14 days
  The distribution of measurement points in each zone was analyzed for A, B, C, D, and E. Zone A is clinically accurate; zone B is clinically uncritical decision; and the remaining zones C, D, and E are inaccurate to varying degrees.
  Analyze the sum of zone A and zone B.
Percentage of total points found in Zone A+B of Consensus Error Grid | From successful device-wearing to device-removal, up to 14 days
  The distribution glucose level points in each zone was analyzed for A, B, C, D, and E. Zone A is no effect on clinical action; zone B is altered clinical action or little or no effect on clinical outcome; Zone C is altered clinical action-likely to affect clinical outcome; and the remaining zones D, E are altered clinical action-could have significant medical risk or dangerous consequences.
  Analyze the sum of zone A and zone B.
Mean absolute relative difference (MARD%) | From successful device-wearing to device-removal, up to 14 days
  MARD% requires an absolute relative difference (ARD) for each subject to be calculated, and then gets the mean for all subjects.

SECONDARY OUTCOMES:
15/15% agreement rate with reference value | From successful device-wearing to device-removal, up to 14 days
  To compare CGM values with reference venous blood glucose values and to analyze the agreement rate
30/30% agreement rate with reference value | From successful device-wearing to device-removal, up to 14 days
  To compare CGM values with reference venous blood glucose values and to analyze the agreement rate
Scores of questionnaire on Ease of Use | Day 14
  A questionnaire on Ease of Use will be used to evaluate the Ease of Use of the study device through user ratings of the study device.
  5-point-scale with 1=Very Unsatisfied, 5=Very Satisfied.
Hyperglycemia or hypoglycemia alarm/alert performance of study device | From successful device-wearing to device-removal, up to 14 days
Number of cases of device failure/defect events | From successful device-wearing to device-removal, up to 14 days
Pain score | Day 1
  The Gracely Box Scale will be used to evaluate the pain level of first CGM sensor insertion, and the pain level of first BGM fingertip blood glucose collection.
  Gracely Box Scale is a visual analog of 0 (0=No pain sensation) to 20, used by a participant to define the pain intensity experience.
Performance of user interfaces or patient interactions: Success rate of sensor insertion, sensor displacement rate, and calibration | From successful device-wearing to planned device-removal, up to 14 days
  Sensor insertion success is defined as the number of sensors used within 10 hours after the first sensor insertion less than or equal to 2.
  Sensor displacement is defined as accidental shedding or displacement of the sensor during wearing.
Number of participants with adverse events/serious adverse events | From day 1 to follow up (day 17 +- 1)
AE with special concern: erythema/edema under the adhesive patch or at the insertion site | From successful device-wearing to device-removal, up to 14 days
  A Draize score (0 to 3) will be used to assess the degree of erythema and edema, with higher scores representing a higher severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Many locations, Multiple Locations, Many Locations
  - Many Locations, Multiple Locations

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — http://clinicaltrials.bayer.com/